CLINICAL TRIAL: NCT03011281
Title: Effectiveness and Safety of Tofacitinib in Korean Patients With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanyang University (Other)
Responsible Party: Principal Investigator, Yoon-Kyoung Sung, Associate professor, Hanyang University
Other Study IDs: HUHRD-SPE-16-09
Record Dates: First submitted 2016-12-30; First posted 2017-01-05 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Hemoglobin Hematocrit WBC Platelet count ESR CRP ALT AST ALP BUN Creatinine Bilirubin Urinalysis Total Cholesterol HDL (Calculated) LDL TG Rheumatoid factor(RF) Anti-nuclear antibodies(ANA) Anti-CCP HbA1c
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA patients who start Tofacitinib: Korean RA patients who start Tofacitinib with moderately to severely active RA who have had an inadequate response or intolerance to methotrexate or biologics.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib
  Other Names: Xeljanz

SUMMARY:
The objectives of this single center, prospective, non-interventional inception cohort is to understand patient characteristics, general treatment patterns, effectiveness, and safety of Tofacitinib for rheumatoid arthritis patients in the real-world setting.

1. To evaluate the baseline characteristics of Korean RA patients treated with Tofacitinib
2. To evaluate the effectiveness and safety of Tofacitinib in clinical practice in Korean RA patients.
3. To further evaluate safety, effectiveness and demographic characteristics of the patients treated with Tofacitinib matched with and compared to biologic DMARDs from the BIOPSY registry database.

ELIGIBILITY:
Inclusion Criteria:

A. Patients who provide a written informed consent form of participating in this study.

B. Patients who are more than 19 years old. C. Patients with moderately to severely active rheumatoid arthritis as defined per EULAR guidelines, who have had an inadequate response or are intolerant to methotrexate.

Exclusion Criteria:

A. Patients who do not provide a written informed consent form of participating in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean RA patients who start Tofacitinib with moderately to severely active RA who have had an inadequate response or intolerance to methotrexate or biologics
Sampling Method: Non-Probability Sample
Enrollment: 378 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
DAS28-ESR (erythrocyte sedimentation rate) remission (DAS28 < 2.6) rate (%) | 5 years

SECONDARY OUTCOMES:
Assessment of efficacy with DAS28 (erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP)) | 5 years
Assessment of safety based on adverse events that occur during 5 years of patient monitoring. | 5 years
Assessment of adherence with Patient-reported Adherence, and Medication Possession Ratio (MPR) at 24, 48, 72, 96, 120, 144, 168, 192, 216 and 240 weeks of clinical visit. | 5 years
Assessment of Quality of life by European Quality of Life-5 Dimensions (EQ-5D) | 5 years
Global Health assessment using Visual Analogue Scale (VAS) | 5 years
Assessment of fatigue by Functional Assessment of Chronic Illness Therapy -Fatigue (FACIT-Fatigue) | 5 years
Assessment of sleep disturbance using Visual Analogue Scale (VAS) | 5 years
Assessment of efficacy with Simple Disease Activity Index (SDAI) | 5 years
Assessment of efficacy with Clinical Disease Activity Index (CDAI) | 5 years
Assessment of efficacy with European League Against Rheumatism (EULAR) response Criteria | 5 years
Assessment of Quality of life by Health Assessment Questionnaire Disability Index (HAQ-DI) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoon-Kyoung Sung, MD, PhD, MPH, Principal Investigator — Hanyang University Hospital for Rheumatic Diseases
Locations (1):
- Hanyang University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No